CLINICAL TRIAL: NCT02525172
Title: Immune Modulation Therapy for ERT-naïve or ERT-treated Pompe Disease Patients
Brief Title: Immune Modulation Therapy for Pompe Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201504036MIPB
Record Dates: First submitted 2015-08-10; First posted 2015-08-17 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Pompe Disease
Keywords: immune modulation therapy; acid α-glucosidase; antibody
MeSH Terms: conditions — Glycogen Storage Disease Type II | interventions — Rituximab; Immunoglobulins, Intravenous; Bortezomib; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ITT (Experimental): immune modulation therapy
  Interventions: Drug: Rituximab; Drug: intravenous immune globulin; Drug: Bortezomib; Drug: Methotrexate

INTERVENTIONS:
Drug: Rituximab
Drug: intravenous immune globulin
Drug: Bortezomib
Drug: Methotrexate

SUMMARY:
The purpose of this study is to assess anti-recombinant human acid α-glucosidase (anti-rhGAA) antibody titers after treatment with immune modulation therapy in patients of Pompe disease.

ELIGIBILITY:
Inclusion Criteria:

* The patient (and/or patient's legal guardian if patient is < 18years) must provide written informed consent prior to any study-related procedures that are performed;
* The patient must have a confirmed diagnosis of Pompe disease defined as a documented acid α-glucosidase (GAA) enzyme deficiency from blood samples or 2 GAA gene mutations;
* The patient (and/or legal guardian) must have ability to comply with clinical protocol;
* Regimen A only: The patient is receiving enzyme replacement therapy, exhibits clinical decline, and has persistent high anti-recombinant human acid α-glucosidase (anti-rhGAA) antibody titers and/or tested positive for antibodies that inhibit enzymatic activity and/or uptake of Myozyme;
* Regimen B only: The patient is cross-reactive immune material (CRIM) -negative AND have not received Myozyme infusion prior to enrollment

Exclusion Criteria:

* The patient is at risk of reactivation or is a carrier of Hepatitis B or Hepatitis C;
* The patient is at risk of reactivation of tuberculosis or has regular contact with individuals who are being actively treated for tuberculosis;
* The patient has used any investigational product (other than alglucosidase alfa) within 30 days prior to study enrollment;
* The patient is pregnant or lactating;
* The patient has had or is required to have any live vaccination within one month prior to enrollment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2015-08; Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
anti-recombinant human acid α-glucosidase (anti-rhGAA) antibody titers decrease | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yin-Hsiu Chien, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Yin-Hsiu Chien, Taipei, Taiwan

REFERENCES:
- [Derived] Chen HA, Hsu RH, Fang CY, Desai AK, Lee NC, Hwu WL, Tsai FJ, Kishnani PS, Chien YH. Optimizing treatment outcomes: immune tolerance induction in Pompe disease patients undergoing enzyme replacement therapy. Front Immunol. 2024 Apr 23;15:1336599. doi: 10.3389/fimmu.2024.1336599. eCollection 2024. PMID 38715621